CLINICAL TRIAL: NCT01110577
Title: Inter-Center Reproducibility Study of Magnetic Resonance Imaging (MRI) for Quantification of Hepatic Fat Fraction in Diabetic and Pre-Diabetic Patients
Brief Title: Study of Magnetic Resonance Imaging (MRI) to Quantify Liver Fat in Diabetic and Pre-Diabetic Patients (0000-171)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-171; 171
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: MRI; Hepatic Steatosis Study
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Traveling cohort: Overweight patients with or without type 2 diabetes or pre-diabetes

SUMMARY:
This study will assess the inter-center reproducibility and accuracy of hepatic fat fraction measurements using up to two MRI-based methods. The intra-class correlation coefficient (ICC) for the repeated measurements is expected to be greater than 0.6.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to travel to MRI centers
* All patients have a BMI ≥27 kg/m2 at the prestudy (screening) visit
* Patient is male or female and at least 18 years of age
* At least 5 patients have type 2 diabetes mellitus or pre-diabetes

Exclusion Criteria:

* Female patient is pregnant or has a positive pregnancy test at screening;
* Patient has known liver disease other than fatty liver
* Patient has a history of neoplastic disease
* Patient is HIV positive
* Patient has known claustrophobia or other contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited for the study
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficient (ICC) for repeated hepatic fat fraction (HFF) measurements from the LIPOQuant method | 28 +/- 7 days from Imaging Visit 1

SECONDARY OUTCOMES:
ICC for repeated HFF measurements from the 3-point Dixon method | 28 +/- 7 days from Imaging Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Mashhood A, Railkar R, Yokoo T, Levin Y, Clark L, Fox-Bosetti S, Middleton MS, Riek J, Kauh E, Dardzinski BJ, Williams D, Sirlin C, Shire NJ. Reproducibility of hepatic fat fraction measurement by magnetic resonance imaging. J Magn Reson Imaging. 2013 Jun;37(6):1359-70. doi: 10.1002/jmri.23928. Epub 2012 Nov 21. PMID 23172799